CLINICAL TRIAL: NCT01033318
Title: A Double-Blind, Double Dummy, Randomized, Placebo-Controlled, Alternating Panel, Single Oral Rising Dose Study to Assess the Pharmacokinetics and Pharmacodynamics of MK1809 in Healthy Young Volunteers
Brief Title: A Study of the Pharmacokinetics and Pharmacodynamics of MK1809 (1809-001)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1809-001; MK1809-001; 2009_703
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (15):
- Part 1 A-1 (Experimental): Part 1; Panel A; Sequence 1:
  2 mg MK1809 / placebo / 50 mg MK1809 / 150 mg MK1809 / 100 mg Losartan
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 1 A-2 (Experimental): Part 1; Panel A; Sequence 2:
  Losartan / 10 mg MK1809 / placebo / 150 mg MK1809 / 280 mg MK1809
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 1 A-3 (Experimental): Part 1; Panel A; Sequence 3 2 mg MK1809 / 10 mg MK1809 / Losartan / Placebo / 280 mg MK1809
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 1 A-4 (Experimental): Part 1; Panel A; Sequence 4 2 mg MK1809 / Losartan / 50 mg MK1809 / 150 mg MK1809 / Placebo
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 1 A-5 (Experimental): Part 1; Panel A; Sequence 5:
  Placebo / 10 mg MK1809 / 50 mg MK1809 / Losartan / 280 mg MK1809
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 1 B-1 (Experimental): Part 1; Panel B; Sequence 1:
  5 mg MK1809 / Placebo / 100 mg MK1809 / 210 mg MK1809 / Placebo with food
  Interventions: Drug: MK1809; Drug: Comparator: Placebo
- Part 1 B-2 (Experimental): Part 1; Panel B; Sequence 2:
  5 mg MK1809 / 25 mg MK1809/ Placebo / Losartan / 25 mg MK1809 with food
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 1 B-3 (Experimental): Part 1; Panel B; Sequence 3:
  5 mg MK1809 / Losartan / 100 mg MK1809 / 210 mg MK1809 / Losartan with food
  Interventions: Drug: MK1809; Drug: Comparator: Losartan
- Part 1 B-4 (Experimental): Part 1; Panel B; Sequence 4:
  Losartan / 25 mg MK1809/ 100 mg MK1809 / Placebo / 25 mg MK1809 with food
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 1 B-5 (Experimental): Part 1; Panel B; Sequence 5:
  Placebo / 25 mg MK1809/ Losartan / 210 mg MK1809 / 25 mg MK1809 with food
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 2 C-1 (Experimental): Part 2; Panel C; Sequence 1:
  50 mg MK1809 / Placebo / 150 mg MK1809 / 210 mg MK1809 / Losartan
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 2 C-2 (Experimental): Part 2; Panel C; Sequence 2:
  50 mg MK1809 / 100 mg MK1809/ Placebo / Losartan / 280 mg MK1809
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 2 C-3 (Experimental): Part 2; Panel C; Sequence 3:
  Losartan / 100 mg MK1809/ 150 mg MK1809 / 210 mg MK1809 / Placebo
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 2 C-4 (Experimental): Part 2; Panel C; Sequence 4:
  50 mg MK1809 / Losartan / 150 mg MK1809 / Placebo / 280 mg MK1809
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo
- Part 2 C-5 (Experimental): Part 2; Panel C; Sequence 5:
  Placebo / 100 mg MK1809/ Losartan / 210 mg MK1809 / 280 mg MK1809
  Interventions: Drug: MK1809; Drug: Comparator: Losartan; Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK1809 — single oral doses of MK1809
Drug: Comparator: Losartan — single oral doses of 100 mg Losartan
  Other Names: Losartan
  Arms: Part 1 A-1; Part 1 A-2; Part 1 A-3; Part 1 A-4; Part 1 A-5; Part 1 B-2; Part 1 B-3; Part 1 B-4; Part 1 B-5; Part 2 C-1; Part 2 C-2; Part 2 C-3; Part 2 C-4; Part 2 C-5
Drug: Comparator: Placebo — Placebo to MK1809
  Arms: Part 1 A-1; Part 1 A-2; Part 1 A-3; Part 1 A-4; Part 1 A-5; Part 1 B-1; Part 1 B-2; Part 1 B-4; Part 1 B-5; Part 2 C-1; Part 2 C-2; Part 2 C-3; Part 2 C-4; Part 2 C-5

SUMMARY:
The goal of this study is to identify at least one safe and well tolerated dose of MK1809 that has similar pharmacokinetic qualities as 100 mg losartan.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Nonsmoker for at least 6 months
* Body Mass Index (BMI) less than or equal to 29 kg/m2
* In overall good health

Part 2:

* Body Mass Index (BMI) greater than 18kg/m2 and less than or equal to 35kg/m2
* In overall good health (patients with hypertension and/or hyperlipidemia are accepted)

Exclusion Criteria:

Part 1:

* History of any cardiovascular disease or any clinically significant family history of cardiac arrhythmias or conduction abnormalities at an age less than 60 years
* History of any major endocrine, vascular, hematologic, gastrointestinal, hepatic, renal or genitourinary disease/disorder
* History of cancer
* Clinically significant history of a neurological disorder (includes epilepsy,stroke, transient ischemic attack, classic migraines)
* Active or history of a psychiatric disorder (includes depression, bipolar disorder, schizophrenia, anxiety)
* History of asthma, severe wheezing, COPD, or other pulmonary disease
* Individual or family history of bleeding or hemorrhagic diathesis, or bleeding difficulties
* Major surgery, donated blood or participated in another investigational drug(s) trial within 30 days
* Illicit drug use (including recreational); or history of drug or alcohol abuse (within 2 years)
* Nitrate therapy within 4 weeks
* History of significant drug allergy or history of food allergies

Part 2

* History of any clinically significant cardiac or cardiovascular disease (other than hypertension)
* History of any major endocrine, vascular, hematologic, gastrointestinal, hepatic, renal or genitourinary disease/disorder
* History of cancer
* History of a neurological disorder (includes epilepsy,stroke, transient ischemic attack, classic migraines)
* Active or history of a psychiatric disorder (includes depression, bipolar disorder, schizophrenia, anxiety)
* History of asthma, severe wheezing, COPD, or other pulmonary disease
* Individual or family history of bleeding or hemorrhagic diathesis, or bleeding difficulties
* Illicit drug use (including recreational); or history of drug or alcohol abuse (within 2 years)
* Surgery, significant blood loss, donated blood, or participated in another investigational drug(s) trial within 30 days
* Nitrate therapy within 4 weeks
* History of significant drug allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09-11 (Actual); Primary Completion 2008-06-19 (Actual); Study Completion 2008-06-19 (Actual)

PRIMARY OUTCOMES:
Part I: Area under the plasma concentration (AUC) versus time curve in healthy adult male subjects in the fasted state | Through 32 hours postdose
Part 1: Trough plasma concentration in healthy adult male subjects in the fasted state | 24 hours postdose
Part 2: Safety and tolerability of rising single oral doses of MK1809 in adult hypertensive patients based on an assessment of clinical and laboratory adverse experiences | Duration of study and up to 14 days after administration of the last dose of study drug

SECONDARY OUTCOMES:
Part 1: Area under the plasma concentration (AUC) versus time curve resulting from a single oral dose of MK1809 following a standard high-fat breakfast (compared to that observed with the identical dose level administered in the fasted state) | 24 hours postdose
Part 1: Maximum concentration of drug in the plasma (Cmax) resulting from a single oral dose of MK1809 following a standard high-fat breakfast (compared to that observed with the identical dose level administered in the fasted state) | Through 32 hours postdose
Part 1: Number of clinical and laboratory adverse experiences (AEs) to assess safety and tolerability | Duration of study and up to 14 days after administration of the last dose of study drug
Part 2: Area under the plasma concentration (AUC) versus time curve of the E3174 metabolite | Through 32 hours postdose
Part 2: Trough plasma concentration of the E3174 metabolite | Through 32 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC